CLINICAL TRIAL: NCT05274269
Title: A Phase 3 Double-blind, Randomized, Placebo-controlled Study Evaluating the Efficacy and Safety of ELX/TEZ/IVA in Cystic Fibrosis Subjects 6 Years of Age and Older With a Non-F508del ELX/TEZ/IVA-responsive CFTR Mutation
Brief Title: Evaluation of Efficacy and Safety of Elexacaftor/Tezacaftor/Ivacaftor (ELX/TEZ/IVA) in Cystic Fibrosis Subjects Without an F508del Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX21-445-124; 2021-005320-38 (EudraCT Number)
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo matched to ELX/TEZ/IVA FDC in the morning and placebo matched to IVA in the evening for 24 weeks.
  Interventions: Other: Placebo (matched to ELX/TEZ/IVA); Other: Placebo (matched to IVA)
- ELX/TEZ/IVA (Experimental): Participants 6 to less than (<) 12 years of age and weighing <30 kilogram (kg) at Day 1 received ELX 100 milligram (mg)/TEZ 50 mg /IVA 75 mg as fixed dose combination (FDC) tablets in the morning and IVA as mono tablet in the evening and those weighing more than or equal to (≥) 30 kg at Day 1 received ELX 200 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 24 weeks. Participants ≥12 years age at Day 1 received ELX 200 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 24 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination (FDC) tablets for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
  Arms: ELX/TEZ/IVA
Drug: IVA — Tablet for oral administration.
  Other Names: VX-770; ivacaftor
  Arms: ELX/TEZ/IVA
Other: Placebo (matched to ELX/TEZ/IVA) — Placebo matched to ELX/TEZ/IVA for oral administration.
  Arms: Placebo
Other: Placebo (matched to IVA) — Placebo matched to IVA for oral administration.
  Arms: Placebo

SUMMARY:
This study evaluated the efficacy, pharmacodynamics (PD) and safety of ELX/TEZ/IVA in participants 6 years of age and older with a non-F508del ELX/TEZ/IVA-responsive cystic fibrosis transmembrane conductance regulator gene (CFTR) mutation.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has a qualifying ELX/TEZ/IVA-responsive CFTR mutation and does not have an exclusionary CFTR mutation
* Forced expiratory volume in 1 second (FEV1) value >=40% and <=100% of predicted mean for age, sex, and height

Key Exclusion Criteria:

* History of solid organ or hematological transplantation
* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 307 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-07-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (90):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Belgium (6):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - Universitair Ziekenhuis Antwerpen (UZA) - Antwerp University Hospital, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert
- Canada (6):
  - Stollery Children's Hospital, Edmonton
  - Centre Hospitalier de l'Universite de Montreal (CHUM) Hotel-Dieu, Montreal
  - McGill University Health Centre, Glen Site, Montreal Children's Hospital, Montreal
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
  - St. Paul's Hospital, Vancouver
- Czechia (2):
  - Klinika Detskych Infekcnich Nemoci, Brno
  - Fakultni nemocnice v Motole, Prague
- France (17):
  - CHU Lyon - Hopital Femme Mere-Enfant, Bron
  - Centre Hospitalier Intercommunal Creteil, Créteil
  - Institut Cœur Poumon, CHU de Lille, Lille
  - CHU Marseille - Hopital Nord, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Centre Hospitalier Universitaire De Nantes - G. R. Laennec, Nantes
  - Centre Hospitalier Universitaire (CHU) de Nice - Hopital Pasteur, Nice
  - Hopital Cochin, Paris
  - Hopital Necker, Enfants Malades, Paris
  - Hopital Robert Debre, Paris
  - Hopital Haut-Leveque - CRCM Adulte, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire De Reims, Hopital Sebastopol, Reims
  - CHU de Rennes - Hôpital Sud, Rennes
  - Centre de Perharidy, Roscoff
  - CHU de Toulouse - Hopital Larre, Toulouse
  - Hopital Bretonneau, Tours
- Germany (19):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitaetsklinkum Koeln, CF-Studienzentrum, Cologne
  - Friedrich-Alexander University of Erlangen-Nuremberg, University Children's Hospital, Erlangen
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Johann Wolfgang Goethe University, Frankfurt
  - Justus-Liebig-Universität Gießen Zentrum für Kinderheilkunde und Jugendmedizin, Giessen
  - Universitätsklinikum Halle (Saale) / Universitätsklinik und Poliklinik für Innere Medizin, Schwerpunkt Pneumologie, Halle
  - Hannover Medical School, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Jena, Mukoviszidose-Zentrum, Jena
  - Johannes Gutenberg-Universitaet, Mainz
  - Dr. von Haunersches Kinderspital, München
  - Klinikum Innenstadt, University of Munich, München
  - Pneumologisches Studienzentrum Muenchen-West, München
  - Klinik fur Kinder- und Jugendmedizin, Universitatsklinikum Munster, Münster
  - Klinikum Westbrandenburg (CF), Potsdam
  - Universitätsklinikum Tübingen Klinik für Kinder- und Jugendmedizin, Tübingen
  - Universitätsklinikum Ulm, Klinik für Kinder- und Jugendmedizin (CF), Ulm
  - Universitätsklinikum Würzburg, Würzburg
- National Koranyi Institute for TBC and Pulmonology, Budapest, Hungary
- Italy (11):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - IRCCS Istituto Giannina Gaslini-Ospedale Pediatrico, Genova
  - Azienda Ospedaliera Universitaria Policlinico G. Martino, Messina
  - Fondazione IRCCS Ospedale Maggiore Policlinico, Mangiagalli e Regina Elena, Milan
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Federico II (Adults), Naples
  - Malattie Apparato Respiratorio 2 - Centro Fibrosi Cistica, Orbassano
  - Centro Regionale Fibrosi Cistica, A.O. Ospedale San Carlo, Potenza
  - Ospedale Pediatrico Bambino Gesu, Rome
  - Azienda Ospedaliera di Verona - Ospedale Civile Maggiore, Verona
- Netherlands (5):
  - Academisch Medisch Centrum (Academic Medical Centre), Amsterdam
  - UMC St. Radboud, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - HagaZiekenhuis van den Haag, The Hague
  - Universitair Medisch Centrum Utrecht, Utrecht
- Oslo University Hospital, Department of Paediatric Medicine, Oslo, Norway
- Poland (3):
  - Pediatric Hospital Polanki named of Maciej Płażyński, Gdansk
  - Institute of Tuberculosis and Lung Diseases, Rabka-Zdrój
  - Instytut Matki i Dziecka, Klinika Mukowiscydozy IMiD, Oddział Chorób Płuc SZPZOZ im.Dzieci Warszawy w Dziekanowie Leśnym, Łomianki
- Portugal (2):
  - Hospital de Santa Maria, Lisbon
  - Hospital Sao Joao, Porto
- Spain (13):
  - Hospital de Cruces, Barakaldo
  - Hospital Saint Joan de Deu, Barcelona
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Infantil La Paz, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Corporacio Sanitaria Parc Tauli - Sabadell Hospital Universitari, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm
- Kinderspital Zuerich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in cystic fibrosis (CF) participants aged 6 years and older with a non-F508del ELX/TEZ/IVA-responsive cystic fibrosis transmembrane conductance regulator gene (CFTR) mutation.
Period: Overall Study
Arm/Group | Placebo | ELX/TEZ/IVA
Started | 102 | 205
Completed | 102 | 197
Not Completed | 0 | 8
Not completed — Adverse Event | 0 | 3
Not completed — Death | 0 | 1
Not completed — Other | 0 | 2
Not completed — Withdrawal of consent (not due to AE) | 0 | 2

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of the study drug were included in the baseline analysis.
Groups:
- ELX/TEZ/IVA: Participants 6 to <12 years of age and weighing <30kg at Day 1 received ELX 100 mg/TEZ 50 mg /IVA 75 mg as FDC tablets in the morning and IVA as mono tablet in the evening and those weighing ≥30 kg at Day 1 received ELX 200 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 24 weeks. Participants ≥12 years age at Day 1 received ELX 200 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | ELX/TEZ/IVA | Total
Number analyzed (Participants) | 102 | 205 | 307
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.9 (16.4) | 33.3 (15.9) | 33.5 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 113 | 165
  Male | 50 | 92 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 88 | 171 | 259
  Not Collected per Local Regulations | 11 | 26 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 86 | 172 | 258
  Asian | 2 | 4 | 6
  Other | 1 | 3 | 4
  Not Collected per Local Regulations | 12 | 26 | 38
  White, Asian | 1 | 0 | 1
Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) [Mean (Standard Deviation); unit: percent predicted FEV1] — FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
  percent predicted FEV1 | 68.1 (18.1) | 67.5 (17.6) | 67.7 (17.7)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Week 24
Population: The Full Analysis Set (FAS) will include all randomized participants who carry the intended mutation and received at least 1 dose of study drug. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted FEV1
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 98 | 192
percent predicted FEV1 | -0.4 [-2.0 to 1.3] | 8.9 [7.7 to 10.0]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Mixed Models for Repeated Measures; LS Mean difference = 9.2, 95% CI 2-sided [7.2 to 11.3]

2. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 24
Population: FAS. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluated for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimole per liter (mmol/L)
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 100 | 200
millimole per liter (mmol/L) | 0.5 [-2.6 to 3.6] | -27.8 [-30.0 to -25.6]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Mixed Models for Repeated Measures; LS Mean difference = -28.3, 95% CI 2-sided [-32.1 to -24.5]

3. Secondary Outcome: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain (RD) Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline Through Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 102 | 202
units on a scale | -2.0 [-5.2 to 1.3] | 17.5 [15.2 to 19.8]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Mixed Models for Repeated Measures; LS Mean difference = 19.5, 95% CI 2-sided [15.5 to 23.5]

4. Secondary Outcome: Absolute Change in Body Mass Index (BMI)
Description: BMI was defined as weight in kilogram (kg) divided by height in square meter (m^2).
Time Frame: From Baseline at Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 102 | 196
kg/m^2 | 0.35 [0.16 to 0.53] | 0.81 [0.68 to 0.94]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Mixed Models for Repeated Measures; LS Mean difference = 0.47, 95% CI 2-sided [0.24 to 0.69]

5. Secondary Outcome: Absolute Change in Weight
Time Frame: From Baseline at Week 24
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kilogram (kg)
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 102 | 196
kilogram (kg) | 1.2 [0.6 to 1.7] | 2.4 [2.1 to 2.8]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p < 0.0001, Mixed Models for Repeated Measures; LS Mean difference = 1.3, 95% CI 2-sided [0.6 to 1.9]

6. Secondary Outcome: Number of Pulmonary Exacerbations (PEx)
Description: Pulmonary exacerbation was defined as the treatment with new or changed antibiotic therapy (intravenous, inhaled, or oral) for greater than or equal to 4 sinopulmonary signs/symptoms.
Time Frame: From Baseline Through Week 24
Population: as for outcome 2
Measure: Number; unit: PEx events
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 102 | 205
PEx events | 40 | 21

7. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 28
Population: Safety Set was defined as all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- ELX/TEZ/IVA: Participants 6 to <12 years of age and weighing <30 kg at Day 1 received ELX 100mg/TEZ 50 mg /IVA 75 mg as FDC tablets in the morning and IVA as mono tablet in the evening and those weighing ≥30 kg at Day 1 received ELX 200 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 24 weeks. Participants ≥12 years age at Day 1 received ELX 200 mg/TEZ 100 mg/IVA 150 mg as FDC tablets in the morning and IVA as mono tablet in the evening for 24 weeks.
Arm/Group | Placebo | ELX/TEZ/IVA
Number analyzed (Participants) | 102 | 205
Participants
  Participants with TEAEs | 97 | 193
  Participants with SAEs | 15 | 18

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 28
Description: Safety Set was defined as all participants who received at least 1 dose of study drug.
Arm/Group | Placebo | ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/102 | 1/205
Serious Adverse Events (participants affected / at risk) | 15/102 | 18/205
Other Adverse Events (participants affected / at risk) | 86/102 | 164/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=102) | ELX/TEZ/IVA (N=205)
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1
Drug intolerance (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 13 | 5
Pneumonia (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=102) | ELX/TEZ/IVA (N=205)
Abdominal pain (Gastrointestinal disorders) | 13 | 17
Abdominal pain upper (Gastrointestinal disorders) | 7 | 10
Constipation (Gastrointestinal disorders) | 4 | 15
Diarrhoea (Gastrointestinal disorders) | 10 | 26
Vomiting (Gastrointestinal disorders) | 7 | 15
Pyrexia (General disorders) | 14 | 27
COVID-19 (Infections and infestations) | 10 | 19
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 36 | 28
Influenza (Infections and infestations) | 2 | 18
Nasopharyngitis (Infections and infestations) | 20 | 42
Rhinitis (Infections and infestations) | 6 | 20
Upper respiratory tract infection (Infections and infestations) | 10 | 17
Headache (Nervous system disorders) | 13 | 37
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 36
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 12
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 17
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 13 | 20
Rash (Skin and subcutaneous tissue disorders) | 1 | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT05274269/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT05274269/SAP_001.pdf